CLINICAL TRIAL: NCT02678962
Title: Comparison of Outcomes With Multifocal Intraocular Lenses
Acronym: COMIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, A-Yong Yu, Clinical Professor, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIOLs2016
Record Dates: First submitted 2016-02-01; First posted 2016-02-10 (Estimated); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Cataract
Keywords: Multifocal Intraocular Lenses; bilateral implantation
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- SN6AD1 group (Active Comparator): Bilateral cataract surgery with implantation of SN6AD1 multifocal IOLs
  Interventions: Device: SN6AD1
- SBL-3 group (Active Comparator): Bilateral cataract surgery with implantation of SBL-3 multifocal IOLs
  Interventions: Device: SBL-3
- LS-313 MF30 group (Active Comparator): Bilateral cataract surgery with implantation of LS-313 MF30 multifocal IOLs
  Interventions: Device: LS-313 MF30
- AT LISA tri 839 MP group (Active Comparator): Bilateral cataract surgery with implantation of AT LISA tri 839 MP multifocal IOLs
  Interventions: Device: AT LISA tri 839 MP
- ART group (Active Comparator): Bilateral cataract surgery with implantation of ART toric multifocal IOLs
  Interventions: Device: ART
- LS-313 MF30T group (Active Comparator): Bilateral cataract surgery with implantation of LS-313 MF30T toric multifocal IOLs
  Interventions: Device: LS-313 MF30T

INTERVENTIONS:
Device: SN6AD1 — Bilateral cataract surgery with implantation of SN6AD1 multifocal IOLs
  Arms: SN6AD1 group
Device: SBL-3 — Bilateral cataract surgery with implantation of SBL-3 multifocal IOLs
  Arms: SBL-3 group
Device: LS-313 MF30 — Bilateral cataract surgery with implantation of LS-313 MF30 multifocal IOLs
  Arms: LS-313 MF30 group
Device: AT LISA tri 839 MP — Bilateral cataract surgery with implantation of AT LISA tri 839 MP multifocal IOLs
  Arms: AT LISA tri 839 MP group
Device: ART — Bilateral cataract surgery with implantation of ART toric multifocal IOLs
  Arms: ART group
Device: LS-313 MF30T — Bilateral cataract surgery with implantation of LS-313 MF30T toric multifocal IOLs
  Arms: LS-313 MF30T group

SUMMARY:
The purpose of this study is to compare and evaluate the clinical outcomes of 6 kinds of Multifocal Intraocular Lenses: SN6AD1, SBL-3, LS-313 MF30, AT LISA tri 839 MP, ART, LS-313 MF30T.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled trial to compare and evaluate the clinical outcomes of 6 kinds of Multifocal Intraocular Lenses, the outcome measurements include postoperative visual acuity, visual quality and complications. Patients enrolled in the study will be randomized to receive one of the Multifocal Intraocular Lenses mentioned above, and the clinical outcomes of each Multifocal Intraocular Lens will be assessed at several visits: 1 day, 1 week, 1 month, 3 months and months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Age from 40 to 80 years old, either gender;
* Patients with bilateral age related cataracts, require bilateral cataract phacoemulsification combined Intraocular Lens implantation;
* Willing to undergo second eye surgery within 7 days after first eye surgery;
* The potential postoperative visual acuity of 20/40 or better in both eyes;
* Preoperative measurement of corneal astigmatism indicate the subjects are suitable for multifocal intraocular lenses implantation;
* Capability to understand the informed consent and willing and able to attend study

Exclusion Criteria:

* Preexisting ocular diseases or conditions other than age related cataracts, have contraindications for cataract surgery;
* Preexisting systemic diseases or conditions that may confound the results of the study;
* Previous ocular surgery history or ocular trauma that may confound the results of the study;
* Require combined surgery that may confound the results of the study;
* Previous participation in other clinical trial within 30 days of this study start;
* Systemic or ocular medications that may confound the outcome of the intervention
* Pregnant, lactating, or planning to become pregnant during the course of the trial;

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-02; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Uncorrected Visual Acuity (UCVA) at Distance, Near | 3 months after surgery
Best distance corrected Visual Acuity at Distance, Near | 3 months after surgery
Defocus curve | 3 months after surgery
  measured with distance correction for unilateral and bilateral
Contrast sensitivity | 3 months after surgery
  measured with CSV-1000HGT(VECTOR VISION, Greenville, OH)
Ocular aberration | 3 months after surgery
  measured with a custom-built aberrometer
Ocular Scatter Index measured by Optical Quality Analysis System(OQAS) II | 3 months after surgery
Modulation Transfer Function (MTF) cut-off measured by OQAS II | 3 months after surgery
Strehl Ratio measured by OQAS II | 3 months after surgery
Quality of Vision (QoV) Questionnaire score | 3 months after surgery
Catquest- 9SF Questionnaire score | 3 months after surgery

SECONDARY OUTCOMES:
Refractive error after surgery | 3 months after surgery
Rate of Posterior Capsule Opacification | 6 months after surgery
Rate of Nd:YAG Laser Posterior Capsulotomy | 6 months after surgery
Rate of Spectacle Independence | 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: AYong Yu, MD. PhD., Principal Investigator — Wenzhou Medical University
Locations (1):
- The Eye Hispital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No